CLINICAL TRIAL: NCT02932800
Title: Fixing the Short Stay Central Venous Catheter: Comparison of Two Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Mário Lúcio Marques Leal, MD, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mario2015
Record Dates: First submitted 2016-09-04; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Suture, Complication
Keywords: Catheters; Vascular Access Devices; Suture Techniques; microbiota; Blood Circulation
MeSH Terms: interventions — CASP8 and FADD-Like Apoptosis Regulating Protein; Culture Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "Ballerina" associated with flap fixation (Active Comparator): The catheter is anchored to the skin begins by a point "U" around the catheter insertion site and followed by a series of woven points around the catheter , commonly referred to as " node dancer " to pass the wires on each side of the orifices located at the catheter distal flaps and hold three consecutive nodes . Then, the clamping is carried out of the catheter to the skin by means of a simple point and hold three consecutive nodes in each lateral hole of the fastening flap while leaving, between the fastening flap and the puncture site a space 2 cm distance for viewing the ostium .
  Interventions: Procedure: Fixation with "ballerina" technique and flip; Other: Evaluation on the third and fift days, filogisticos and infectious signs, fixing loss, and culture
- the usual fixation technique (Active Comparator): The catheter is attached to the skin with a simple point and holding three we row on each side hole fixing fin while leaving, between the fastening flap and the puncture site , an area of 2 cm away for viewing ostium . The catheter is anchored to the skin by a simple point and holding three consecutive us in each hole of the side flap in the distal region.
  Interventions: Procedure: Habitual Fixation; Other: Evaluation on the third and fift days, filogisticos and infectious signs, fixing loss, and culture

INTERVENTIONS:
Procedure: Fixation with "ballerina" technique and flip
  Arms: "Ballerina" associated with flap fixation
Procedure: Habitual Fixation — Evaluation on the third and fift days, filogisticos and infectious signs, fixing loss, and culture
  Arms: the usual fixation technique
Other: Evaluation on the third and fift days, filogisticos and infectious signs, fixing loss, and culture

SUMMARY:
Context: The central venous catheter is used in intensive care units for several indications, including the administration of drugs with sclerosis potential, infusion solutions and hemodynamic monitoring. It can be accessed by per cutaneous puncture using the Seldinger technique, which is an extremely common procedure in intensive care units. The displacement or accidental removal of central venous catheter caused by poor fixation have received little attention, but imply potentially life threatening caused by the complications which can result from the removal of the catheter and the need for reinsertion. Among these complications, can mention the interruption of vital therapies (inotropic and vasopressor drugs) and hemorrhagic shock. In fixing the catheter, the literature is not sufficient to assess whether sutures, staples or tapes are associated with a higher risk of infections. Objective: To compare the efficiency in fixing the short stay central venous catheter using the "Ballerina" technique associated with flap fixation to the usual fixation technique and to observe differences in colonization of microorganisms on the device insertion site. Methods: The investigators propose an individual study, analytical, intervention, longitudinal, prospective, controlled clinical trial and randomized to be developed in the Intensive Care Unit Adult Clinical and Surgical of The Samuel Libânio Clinical Hospital in The University of Sapucaí Valley and Intensive Care Unit Adult Clinical and Surgical of The Hospital e Maternity Santa Paula. After admission of the patient in the Intensive Care Unit and obtaining informed consent and informed, with indication of the short stay central venous catheter, the patient will be allocated through a table of random numbers for the groups: Habitual Fixation (n = 31) and Fixation with "ballerina" technique and flip (n = 31). The participants will evaluate fixation efficiency and colonization of the device's insertion site.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for the use of central venous catheters ;
* Both genders ;
* Age greater than 18 years;
* Admitted to the intensive care unit;
* Informed Consent signed ( by the patient or family ) ;

Exclusion Criteria:

* Device repositioning Need for abnormal pathway or malposition after installation;
* No more indication of the central venous catheter use before the minimum period of 03 days ;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes in catheter fixation | The evaluation will be on the third and fifth day after implantation
  traction, kicking off, fixing loss of the device

OTHER OUTCOMES:
Skin evaluation | The evaluation will be on the third and fifth day after implantation
  It will be evaluation, the presence of hyperemia or not
Local Culture | Will be collected a local swab at the third and fifth day after implantation.
  The material will be seed at least 6 hours, and analyzed after 48h incubation

CONTACTS AND LOCATIONS:
Locations (1):
- Mario Lucio Leal, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided